CLINICAL TRIAL: NCT03566056
Title: Early Recovery Outcomes After Standardized Fast-track Whipples Procedure
Status: Completed | Type: Observational
Sponsor: Eske Kvanner Aasvang (Other)
Responsible Party: Sponsor-Investigator, Eske Kvanner Aasvang, Principle investigator, Associate professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: RH-2016-304-potawhipple
Record Dates: First submitted 2018-04-10; First posted 2018-06-21 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Complications to Whipples procedure — Patients undergoing the Whipple procedure often tend to have a lot of complications. This study aims to investigate what complications these patients experience

SUMMARY:
Today the Whipple procedure is the preferred operation for malignancy in the pancreas. In abdominal surgery this procedure is known for its high surgical stress-response in the patient, which has been attempted to be resolved with the introduction of preoperative high-dose steroids and goal-directed fluid therapy (GDT). Despite this effort, complications still occur regularly (30%) in the first weeks after the operation here at Rigshospitalet. Therefore there is still a challenge in the patients who have undergone the Whipple procedure in the acute postoperative phase. This shows in for example at Rigshospitalet, where 50% of the patients continue to be in the need of vasoactive medication the morning after the operation.

Nevertheless, no studies have in detail described the acute (<24h) postoperative phase. There is also an importance in the fact that there is often no description or control over other important factors, for example medicine with influence on the circulatory system, fluid treatment and response to this etc..

The purpose of this study is to investigate what issues or complications, in particular those of circulatory matter that occurs in this particular group of patients 24 hours after the operation. Furthermore there is lacking a description of which cause-response- link there can be between early and later (30 days) complications, as well as when each of these complications occur. Therefore, there will also be collected data on complications within the first 30 days after the operation for the purpose of a later secondary publication with the same authors.

ELIGIBILITY:
Inclusion Criteria:

* the patient has undergone the Whipple procedure
* The patient is over 18 years ol
* The patient has signed a consent statement from the postoperative therapy ward

Exclusion Criteria:

* The patient did not receive 125 mg of methylprednisolone prior to the operation
* The patient did only undergo pancreatectomy
* The patient wasn't given epidural anesthesia
* the patient was given anesthesia through a mask

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients included is chosen from all the patients in the surgery ward when they have undergone the Whipples procedure and furthermore meet the criteria listed above.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2018-07-18 (Actual); Study Completion 2018-07-18 (Actual)

PRIMARY OUTCOMES:
Hypotension, defined as mean arterial bloodpressure <65 mmHg, measured by invasive arterial blood-pressure, the first morning after surgery at 06.00 (AM) | 6 am on the day after surgery
  Number of patients with the need for nor-adrenalin infusion to maintain mean arterial blood-pressure >65 mmHg, the first morning after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
This has jet not been discussed within the group